CLINICAL TRIAL: NCT04800146
Title: A Prospective Observational Study on the Immune-response to SARS-CoV-2 Vaccination in Cancer Patients - the IOSI-COVID-19-001 Study
Brief Title: A Study on the Immune-response to COVID-19 Vaccination in Cancer Patients - the IOSI-COVID-19-001 Study
Status: Completed | Type: Observational
Sponsor: Ilaria Colombo (Other)
Collaborators: Institute for Research in Biomedicine (Unknown); Ente Ospedaliero Cantonale, Bellinzona (Other)
Responsible Party: Sponsor-Investigator, Ilaria Colombo, Principal Investigator, Oncology Institute of Southern Switzerland
Organization: Oncology Institute of Southern Switzerland (Other)
Other Study IDs: IOSI-COVID19-001
Record Dates: First submitted 2021-03-10; First posted 2021-03-16 (Actual); Last update posted 2023-03-23 (Actual); Status verified 2023-03

CONDITIONS: Covid19; Cancer
MeSH Terms: conditions — COVID-19; Neoplasms | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (8):
- Cohort 1: patients with solid tumors treated with chemotherapy (ongoing or completed no more than 6 months before enrollment). Specific type of chemotherapy inducing similar immunosuppression will be selected (including but not limited to platinum-based combinations, anthracycline combinations, triweekly docetaxel).
  Interventions: Procedure: Blood sample
- Cohort 2: patients with solid tumors treated with single agent immune-check points inhibitors (ongoing or completed no more than 6 months before the enrollment
  Interventions: Procedure: Blood sample
- Cohort 3: patients with solid tumors treated with hormonal agents (ongoing or completed no more than 6 months before enrollment): any anti-androgen for prostate cancer and any anti-estrogen for breast cancer patients.
  Interventions: Procedure: Blood sample
- Cohort 4: patients with previously untreated mature B cell tumors in watch and wait
  Interventions: Procedure: Blood sample
- Cohort 5: patients with mature B cell tumors treated with anti-CD20 monoclonal antibody either alone or in combination with chemotherapy (ongoing or completed no more than 12 months before enrollment
  Interventions: Procedure: Blood sample
- Cohort 6: patients with hematological malignancies treated with pathway inhibitors (ongoing or completed no more than 12 months before enrollment). Different type of targeted agents can be considered, including Bruton tyrosine kinase (BTK) inhibitors, B-cell lymphoma 2 (BCL-2) inhibitors or phosphoinositide-3 kinase (PI3K) inhibitors
  Interventions: Procedure: Blood sample
- Cohort 7: patients with hematological malignancies who have received autologous stem cell or allogenic transplant within 12 months
  Interventions: Procedure: Blood sample
- Cohort 8: non-cancer subjects (age and gender matched) referred to the Division of Infectious Diseases, Lugano, EOC for vaccination against SARS-CoV-2.
  Interventions: Procedure: Blood sample

INTERVENTIONS:
Procedure: Blood sample — Patients will be asked to provide blood samples at specified time points: before and after the SARS-CoV-2 vaccination

SUMMARY:
This is a single centre prospective observational study to assess the immune response to SARS-CoV-2 vaccines in cancer patients receiving active treatment or in follow-up at the IOSI and in non-cancer patients (age and gender matched).

DETAILED DESCRIPTION:
This study will be conducted on 7 cohorts of cancer patients and 1 cohort of non-cancer subjects (age and gender matched) with a sample size of 30 patients in each cohort:

All enrolled patients will be asked to provide blood samples (2 x 10cc Heparin Tubes) at the following time points:

* Baseline: before the administration of the first dose of the SARS-CoV-2 vaccine (within 4 weeks).
* Before the second dose of the SARS-CoV-2 vaccine (within 7 days).
* Follow-up: after 3, 6, 9 and 12 months after the second dose of the SARS-CoV-2 vaccine. A +/- 14 days window is allowed at each follow-up time point.

ELIGIBILITY:
Inclusion Criteria:

* Male of Female age at least 18 years
* Patients with a diagnosis of malignancy (solid tumors or hematological malignancies) according to the defined cohorts. Only for cohorts 1-7
* Eastern Cooperative Oncology Group (ECOG) Performance Status 0-2
* Absence of known immune deficiency (other than cancer for cohorts 1-7)
* Ability to understand the patient information and study consent. Signed and dated written informed consent must be available before performing any study-related procedure
* Willing and able to comply with the study procedures.
* Willing to receive an mRNA anti-SARS-CoV-2 vaccine.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: The population of this study is represented by patients with a diagnosis of solid tumor or hematological malignancy and receiving treatment or on active surveillance at the IOSI who have planned to receive an mRNA (messenger ribonucleic acid) SARS-CoV-2 vaccine, according to the prespecified cohorts.
  A control group of non-cancer subjects followed at the outpatient clinic of the Division of Infectious Diseases, EOC will also be enrolled for comparative analysis.
Sampling Method: Non-Probability Sample
Enrollment: 177 (Actual)
Dates: Start 2021-02-25 (Actual); Primary Completion 2023-03-21 (Actual); Study Completion 2023-03-21 (Actual)

PRIMARY OUTCOMES:
Immune response to SARS-CoV-2 vaccine in cancer patients | 3, 6, 9 and 12 months following vaccination
  to determine the changes in the titer of serum antibodies (IgM, IgG and IgA) targeting SARS-CoV-2 antigens in 7 cohorts of cancer patients who have received the SARS-CoV-2 vaccination. A cohort of non-cancer subjects will be used as control group.

SECONDARY OUTCOMES:
changes in serum antibodies anti SARS-CoV-2 after vaccination | 3, 6, 9 and 12 months following vaccination
  To explore the dynamic changes overtime of the levels of antibodies against SARS-CoV-2 following vaccination in cancer patients and controls
Cellular immune response to SARS-CoV-2 vaccine | 3, 6, 9 and 12 months following vaccination
  To explore the dynamic changes overtime of the T cells immune response following SARS-CoV-2 vaccination in cancer patients and controls.
Cellular immune response to SARS-CoV-2 vaccine | 3, 6, 9 and 12 months following vaccination
  To explore the dynamic changes overtime of the B cells immune response following SARS-CoV-2 vaccination in cancer patients and controls.
Immune response to SARS-CoV-2 vaccine according tumor and treatment type | 3, 6, 9 and 12 months following vaccination
  To explore the correlation between the immune response against SARS-CoV-2 vaccination and the type of cancer (e.g., solid tumors versus hematological malignancies) and the type of anticancer treatment (e.g., anti-CD20, chemotherapy, targeted agents, immunotherapy, allogenic or autologous transplant)

CONTACTS AND LOCATIONS:
Locations (1):
- Oncology Institute of Southern Switzerland, Bellinzona, Switzerland

IPD SHARING:
Plan to Share IPD: No